CLINICAL TRIAL: NCT06817512
Title: Health Effects of Vitamin K2 Supplementation on Skeletal Muscle and Neurological Function After Ischemic Stroke
Brief Title: Ischemic Stroke Nutrition Intervention Study
Acronym: ISNIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Ying Li, Professor, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMUIRB2024027
Record Dates: First submitted 2025-01-14; First posted 2025-02-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke
Keywords: Vitamin K2; Skeletal Muscle; Neurological Function; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K2 (Experimental): Vitamin K2 (menaquinone-7), 300µg/d, one capsule per day
  Interventions: Dietary Supplement: Vitamin K2
- Placebo Control (Placebo Comparator): Placebo with similar appearance and taste, one capsule per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — Vitamin K2 (MK-7) 300µg/d for 1 year
  Arms: Vitamin K2
Dietary Supplement: Placebo — Placebo for 1 year
  Arms: Placebo Control

SUMMARY:
The primary goal of this clinical trial is to assess whether vitamin K2 supplementation can effectively improve skeletal muscle and neurological function in patients with ischemic stroke. The main questions it aims to answer are: 1. Does supplementation with vitamin K2 improve the subjects' muscle strength and muscle mass? 2. Can supplementation with vitamin K2 improve the subjects' neurological function after a stroke? Researchers will compare vitamin K2 supplements with a placebo to observe whether vitamin K2 supplementation can improve skeletal muscle and neurological function in patients with ischemic stroke. Participants will: 1. Take vitamin K2 (MK-7) or a placebo daily for 1 year. 2. Attend face-to-face visits and provide biological samples and relevant data at 0, 3, 6, and 12 months. At 9 months, the visit will be online. After the intervention, follow-up will continue for 1 year to observe the long-term effects.

ELIGIBILITY:
Inclusion Criteria：

Participants who meet all the following conditions will be included in the trial:

1. Men or women aged ≥ 18 years.
2. Patients with recent ischemic stroke（first or recurrent stroke no more than 7 days before admission）without significant residual limb paralysis, NIHSS score between 2-15, and muscle strength graded 2-4.
3. The patient and their legal guardian (or legally acceptable representative) voluntarily sign the informed consent form.

Exclusion Criteria：

Participants who meet any of the following conditions will be excluded from the trial:

1. Presence of consciousness disorders, aphasia, or swallowing disorders.
2. The diagnosis or suspicion of cerebral hemorrhage, atrial fibrillation, or other factors leading to cardiogenic cerebral infarction.
3. Coagulation dysfunction or use of vitamin K antagonists.
4. Suffering from chronic gastrointestinal malabsorption (such as celiac disease, short bowel syndrome), severe congestive heart failure, malignant hypertension, severe liver and kidney dysfunction, persistent malignant tumors (continuous treatment, or diagnosis of malignant tumors<5 years), or other related diseases considered by researchers that seriously affect the patient's survival.
5. Having musculoskeletal diseases or cognitive impairment before the stroke.
6. Currently using or planning to use non research approved dietary supplements during the study period.
7. Currently using or planning to use drugs that affect cognitive or neurological function during the research period.
8. Restricted normal eating or currently receiving enteral or parenteral nutrition support.
9. Contraindications for MRI and other examinations.
10. Currently pregnant or planning pregnancy, currently breastfeeding.
11. Participated in a clinical trial using experimental drugs or devices within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2025-03-23 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Handgrip strength was measured in participants using an electronic dynamometer.

SECONDARY OUTCOMES:
Sustained effects of the intervention on handgrip strength | Measurements were recorded at 24 months (end of follow-up).
  The change in handgrip strength from month 12 (end of intervention) to month 24 (end of follow-up) was assessed. This evaluation aimed to determine the sustained impact of the intervention on handgrip strength following the discontinuation of treatment.
National Institute of Health Stroke Scale (NIHSS) score | Measurements were taken at 0 (baseline), 3, 6, 9, 12 (end of intervention), and 24 (end of follow-up) months.
  The severity of neurological deficits in participants was evaluated using the National Institutes of Health Stroke Scale (NIHSS). This scale provides a standardized assessment, with total scores ranging from 0 (indicating no deficit) to 42 (representing severe neurological injury).
Modified Rankin Scale (mRS) score | Measurements were taken at 0 (baseline), 3, 6, 9, 12 (end of intervention), and 24 (end of follow-up) months.
  The functional neurological recovery of participants will be assessed using the Modified Rankin Scale (mRS). This scale (0-6) quantifies post-stroke disability, where lower scores indicate better outcomes.
Mini-Mental State Examination (MMSE) score | Measurements were taken at 0 (baseline), 3, 6, 9, 12 (end of intervention), and 24 (end of follow-up) months.
  The Mini-Mental State Examination (MMSE) will be administered to patients to evaluate cognitive function across multiple domains using a validated 30-point scale (0, severe impairment; 30, intact cognition), with higher scores indicating better cognitive performance.
Change in ischemic lesion volume | Measurements were taken at 0 (baseline) and 12 (end of intervention) months.
  This study will assess changes in head MRI of patients with ischemic stroke. Change in ischemic lesion volume includes enlargement or reduction of infarcts and the appearance of new ischemic lesions.
Change in white matter lesions | Measurements were taken at 0 (baseline) and 12 (end of intervention) months.
  The progression of white matter lesions (especially in high-signal white matter and lesion expansion) will be detected through head MRI.
Change in cerebral blood flow and function | Measurements were taken at 0 (baseline) and 12 (end of intervention) months.
  Cerebral blood flow and function (arterial blood supply and other ischemia-related imaging features) will be detected through head MRI.
Change in overall brain structural | Measurements were taken at 0 (baseline) and 12 (end of intervention) months.
  The overall brain structural changes (brain atrophy and ventricular enlargement) will be detected through head MRI.
Body composition | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
  The body composition of patients will be measured using bioelectrical impedance analysis (BIA).
Fugl-Meyer Assessment (FMA) score | Measurements were taken at 0 (baseline), 3, 6,12 (end of intervention), and 24 (end of follow-up) months.
  The Fugl-Meyer Assessment (FMA) was employed to evaluate motor function in the patient's upper and lower limbs, with total scores ranging from 0 to 100, where higher scores indicate better motor recovery.
Functional lower extremity strength | Measurements were taken at 0 (baseline), 3, 6,12 (end of intervention), and 24 (end of follow-up) months.
  The functional lower extremity strength of patients will be evaluated through the 30-second Chair Stand Test (CST).
Gait performance | Measurements were taken at 0 (baseline), 3, 6,12 (end of intervention), and 24 (end of follow-up) months.
  The gait performance of patients will be measured using 6-meter walk tests.
Carotid intima-media thickness (IMT) | Measurements were taken at 0 (baseline),6, and 12 (end of intervention) months.
  The patients will receive carotid artery ultrasonography to quantify carotid intima-media thickness (IMT).
Carotid plaques | Measurements were taken at 0 (baseline),6, and 12 (end of intervention) months.
  The patients will undergo carotid artery ultrasonography to detect changes in carotid plaques.
Brachial-ankle PWV (baPWV) | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Ankle Brachial Index (ABI) | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Body weight | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Waist circumference | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Hip circumference | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Upper arm circumference | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Thigh circumference | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Calf circumference | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Blood pressure (systolic pressure and diastolic pressure) | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Heart rate | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
Hospital Anxiety and Depression Scale (HADS） | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
  The Hospital Anxiety and Depression Scale (HADS) was administered to the patients, with the anxiety (HADS-A) and depression (HADS-D) subscales each yielding scores from 0 (asymptomatic) to 21 (severe symptoms).
Pittsburgh Sleep Quality Index (PSQI) | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
  The sleep quality of each patient will be evaluated by the Pittsburgh Sleep Quality Index (PSQI), with scores ranging from 0 to 21, with higher scores indicating poorer sleep quality
Life quality | Measurements were taken at 0 (baseline), 3, 6, 12 (end of intervention), and 24 (end of follow-up) months.
  The SF-36 assesses 8 health domains (physical or mental function, pain, vitality, etc.) through 36 Likert-scale questions. Scores range from 0 (worst health) to 100 (best health) per domain.
Vitamin K2-related biomarkers | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Blood samples from the patients will be tested for biomarkers related to vitamin K2 (e.g., serum vitamin K2, dephosphorylated uncarboxylated matrix Gla-protein (dp-ucMGP)).
Glycemic parameters | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Blood samples from the patients will be tested for glycemic parameters (e.g., fasting blood glucose, fasting insulin).
Lipid metabolism parameters | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Blood samples from the patients will be tested for lipid metabolism parameters (e.g., serum total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C)).
Inflammation-related indicators | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Blood samples from the patients will be tested for inflammation-related markers (e.g., IL-1β, IL-6, IL-8, IL-10, TNF-α, TGF-β, TNF-α-induced protein 3 (TNFAIP3), C-reactive protein (CRP)).
Muscle damage and cardiovascular health-related indicators | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Blood samples from the patients will be tested for muscle damage and cardiovascular health indicators (e.g., creatine kinase (CK) and myoglobin (Mb)).
Blood transcriptomics | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Transcriptomic sequencing will be performed on blood samples collected from the patients to observe changes in blood transcriptional levels.
Metabolomics in serum, urine, and feces | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Metabolomic sequencing will be performed on serum, urine, and fecal samples collected from the patients to observe changes in metabolic levels.
Gut and oral microbiome | Measurements were taken at 0 (baseline), 3, 6, and 12 (end of intervention) months.
  Microbiome sequencing will be conducted on fecal and saliva samples collected from the patients.
Occurrence of cardiovascular and cerebrovascular events | Measurements were taken at 3, 6, 9, 12 (end of intervention), and 24 (end of follow-up) months.
  Cardiovascular and cerebrovascular events of the patients will be monitored during the follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hongqi Hospital Affiliated to Mudanjiang Medical University, Mudanjiang, Heilongjiang
  - The Second Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohsaki Y, Shirakawa H, Miura A, Giriwono PE, Sato S, Ohashi A, Iribe M, Goto T, Komai M. Vitamin K suppresses the lipopolysaccharide-induced expression of inflammatory cytokines in cultured macrophage-like cells via the inhibition of the activation of nuclear factor kappaB through the repression of IKKalpha/beta phosphorylation. J Nutr Biochem. 2010 Nov;21(11):1120-6. doi: 10.1016/j.jnutbio.2009.09.011. Epub 2010 Feb 9. PMID 20149620
- [Background] Tsang CK, Kamei Y. Novel effect of vitamin K(1) (phylloquinone) and vitamin K(2) (menaquinone) on promoting nerve growth factor-mediated neurite outgrowth from PC12D cells. Neurosci Lett. 2002 Apr 19;323(1):9-12. doi: 10.1016/s0304-3940(01)02550-2. PMID 11911978
- [Background] Gely-Pernot A, Coronas V, Harnois T, Prestoz L, Mandairon N, Didier A, Berjeaud JM, Monvoisin A, Bourmeyster N, De Frutos PG, Philippe M, Benzakour O. An endogenous vitamin K-dependent mechanism regulates cell proliferation in the brain subventricular stem cell niche. Stem Cells. 2012 Apr;30(4):719-31. doi: 10.1002/stem.1045. PMID 22290807
- [Background] Zhong Z, Wang Y, Guo H, Sagare A, Fernandez JA, Bell RD, Barrett TM, Griffin JH, Freeman RS, Zlokovic BV. Protein S protects neurons from excitotoxic injury by activating the TAM receptor Tyro3-phosphatidylinositol 3-kinase-Akt pathway through its sex hormone-binding globulin-like region. J Neurosci. 2010 Nov 17;30(46):15521-34. doi: 10.1523/JNEUROSCI.4437-10.2010. PMID 21084607
- [Background] Shibata M, Kumar SR, Amar A, Fernandez JA, Hofman F, Griffin JH, Zlokovic BV. Anti-inflammatory, antithrombotic, and neuroprotective effects of activated protein C in a murine model of focal ischemic stroke. Circulation. 2001 Apr 3;103(13):1799-805. doi: 10.1161/01.cir.103.13.1799. PMID 11282913
- [Background] Carrie I, Belanger E, Portoukalian J, Rochford J, Ferland G. Lifelong low-phylloquinone intake is associated with cognitive impairments in old rats. J Nutr. 2011 Aug;141(8):1495-501. doi: 10.3945/jn.110.137638. Epub 2011 Jun 8. PMID 21653572
- [Background] Carrie I, Portoukalian J, Vicaretti R, Rochford J, Potvin S, Ferland G. Menaquinone-4 concentration is correlated with sphingolipid concentrations in rat brain. J Nutr. 2004 Jan;134(1):167-72. doi: 10.1093/jn/134.1.167. PMID 14704312
- [Background] Viegas CS, Rafael MS, Enriquez JL, Teixeira A, Vitorino R, Luis IM, Costa RM, Santos S, Cavaco S, Neves J, Macedo AL, Willems BA, Vermeer C, Simes DC. Gla-rich protein acts as a calcification inhibitor in the human cardiovascular system. Arterioscler Thromb Vasc Biol. 2015 Feb;35(2):399-408. doi: 10.1161/ATVBAHA.114.304823. Epub 2014 Dec 23. PMID 25538207
- [Background] Harshman SG, Shea MK. The Role of Vitamin K in Chronic Aging Diseases: Inflammation, Cardiovascular Disease, and Osteoarthritis. Curr Nutr Rep. 2016 Jun;5(2):90-98. doi: 10.1007/s13668-016-0162-x. Epub 2016 Mar 31. PMID 27648390
- [Background] Lees JS, Chapman FA, Witham MD, Jardine AG, Mark PB. Vitamin K status, supplementation and vascular disease: a systematic review and meta-analysis. Heart. 2019 Jun;105(12):938-945. doi: 10.1136/heartjnl-2018-313955. Epub 2018 Dec 4. PMID 30514729
- [Background] Ronning SB, Pedersen ME, Berg RS, Kirkhus B, Rodbotten R. Vitamin K2 improves proliferation and migration of bovine skeletal muscle cells in vitro. PLoS One. 2018 Apr 4;13(4):e0195432. doi: 10.1371/journal.pone.0195432. eCollection 2018. PMID 29617432
- [Background] Mladenka P, Macakova K, Kujovska Krcmova L, Javorska L, Mrstna K, Carazo A, Protti M, Remiao F, Novakova L; OEMONOM researchers and collaborators. Vitamin K - sources, physiological role, kinetics, deficiency, detection, therapeutic use, and toxicity. Nutr Rev. 2022 Mar 10;80(4):677-698. doi: 10.1093/nutrit/nuab061. PMID 34472618
- [Background] Freeman AM, Morris PB, Barnard N, Esselstyn CB, Ros E, Agatston A, Devries S, O'Keefe J, Miller M, Ornish D, Williams K, Kris-Etherton P. Trending Cardiovascular Nutrition Controversies. J Am Coll Cardiol. 2017 Mar 7;69(9):1172-1187. doi: 10.1016/j.jacc.2016.10.086. PMID 28254181
- [Background] Droujinine IA, Meyer AS, Wang D, Udeshi ND, Hu Y, Rocco D, McMahon JA, Yang R, Guo J, Mu L, Carey DK, Svinkina T, Zeng R, Branon T, Tabatabai A, Bosch JA, Asara JM, Ting AY, Carr SA, McMahon AP, Perrimon N. Proteomics of protein trafficking by in vivo tissue-specific labeling. Nat Commun. 2021 Apr 22;12(1):2382. doi: 10.1038/s41467-021-22599-x. PMID 33888706
- [Background] de Freitas GB, Lourenco MV, De Felice FG. Protective actions of exercise-related FNDC5/Irisin in memory and Alzheimer's disease. J Neurochem. 2020 Dec;155(6):602-611. doi: 10.1111/jnc.15039. Epub 2020 Jun 2. PMID 32396989
- [Background] Febbraio MA, Pedersen BK. Who would have thought - myokines two decades on. Nat Rev Endocrinol. 2020 Nov;16(11):619-620. doi: 10.1038/s41574-020-00408-7. No abstract available. PMID 32839577
- [Background] Sun Y, Zehr EP. Training-Induced Neural Plasticity and Strength Are Amplified After Stroke. Exerc Sport Sci Rev. 2019 Oct;47(4):223-229. doi: 10.1249/JES.0000000000000199. PMID 31283528
- [Background] Park JG, Lee KW, Kim SB, Lee JH, Kim YH. Effect of Decreased Skeletal Muscle Index and Hand Grip Strength on Functional Recovery in Subacute Ambulatory Stroke Patients. Ann Rehabil Med. 2019 Oct;43(5):535-543. doi: 10.5535/arm.2019.43.5.535. Epub 2019 Oct 31. PMID 31693843
- [Background] Jones TA. Motor compensation and its effects on neural reorganization after stroke. Nat Rev Neurosci. 2017 May;18(5):267-280. doi: 10.1038/nrn.2017.26. Epub 2017 Mar 23. PMID 28331232
- [Background] Madureira S, Guerreiro M, Ferro JM. Dementia and cognitive impairment three months after stroke. Eur J Neurol. 2001 Nov;8(6):621-7. doi: 10.1046/j.1468-1331.2001.00332.x. PMID 11784347
- [Background] Guo J, Wang J, Sun W, Liu X. The advances of post-stroke depression: 2021 update. J Neurol. 2022 Mar;269(3):1236-1249. doi: 10.1007/s00415-021-10597-4. Epub 2021 May 30. PMID 34052887
- [Background] Wechsler LR, Adeoye O, Alemseged F, Bahr-Hosseini M, Deljkich E, Favilla C, Fisher M, Grotta J, Hill MD, Kamel H, Khatri P, Lyden P, Mirza M, Nguyen TN, Samaniego E, Schwamm L, Selim M, Silva G, Yavagal DR, Yenari MA, Zachrison KS, Boltze J, Yaghi S; XIIth Stroke Treatment Academic Industry Roundtable. Most Promising Approaches to Improve Stroke Outcomes: The Stroke Treatment Academic Industry Roundtable XII Workshop. Stroke. 2023 Dec;54(12):3202-3213. doi: 10.1161/STROKEAHA.123.044279. Epub 2023 Oct 27. PMID 37886850
- [Background] Tu WJ, Zhao Z, Yin P, Cao L, Zeng J, Chen H, Fan D, Fang Q, Gao P, Gu Y, Tan G, Han J, He L, Hu B, Hua Y, Kang D, Li H, Liu J, Liu Y, Lou M, Luo B, Pan S, Peng B, Ren L, Wang L, Wu J, Xu Y, Xu Y, Yang Y, Zhang M, Zhang S, Zhu L, Zhu Y, Li Z, Chu L, An X, Wang L, Yin M, Li M, Yin L, Yan W, Li C, Tang J, Zhou M, Wang L. Estimated Burden of Stroke in China in 2020. JAMA Netw Open. 2023 Mar 1;6(3):e231455. doi: 10.1001/jamanetworkopen.2023.1455. PMID 36862407
- [Background] Hu S, Cui B, Mlynash M, Zhang X, Mehta KM, Lansberg MG. Stroke epidemiology and stroke policies in China from 1980 to 2017: A systematic review and meta-analysis. Int J Stroke. 2020 Jan;15(1):18-28. doi: 10.1177/1747493019873562. Epub 2019 Sep 22. PMID 31543073
- [Background] Wang YJ, Li ZX, Gu HQ, Zhai Y, Zhou Q, Jiang Y, Zhao XQ, Wang YL, Yang X, Wang CJ, Meng X, Li H, Liu LP, Jing J, Wu J, Xu AD, Dong Q, Wang D, Wang WZ, Ma XD, Zhao JZ; China Stroke Statistics Writing Committee. China Stroke Statistics: an update on the 2019 report from the National Center for Healthcare Quality Management in Neurological Diseases, China National Clinical Research Center for Neurological Diseases, the Chinese Stroke Association, National Center for Chronic and Non-communicable Disease Control and Prevention, Chinese Center for Disease Control and Prevention and Institute for Global Neuroscience and Stroke Collaborations. Stroke Vasc Neurol. 2022 Oct;7(5):415-450. doi: 10.1136/svn-2021-001374. Epub 2022 Apr 20. PMID 35443985
- [Background] Wang L, Zhou B, Zhao Z, Yang L, Zhang M, Jiang Y, Li Y, Zhou M, Wang L, Huang Z, Zhang X, Zhao L, Yu D, Li C, Ezzati M, Chen Z, Wu J, Ding G, Li X. Body-mass index and obesity in urban and rural China: findings from consecutive nationally representative surveys during 2004-18. Lancet. 2021 Jul 3;398(10294):53-63. doi: 10.1016/S0140-6736(21)00798-4. PMID 34217401
- [Background] Wang L, Peng W, Zhao Z, Zhang M, Shi Z, Song Z, Zhang X, Li C, Huang Z, Sun X, Wang L, Zhou M, Wu J, Wang Y. Prevalence and Treatment of Diabetes in China, 2013-2018. JAMA. 2021 Dec 28;326(24):2498-2506. doi: 10.1001/jama.2021.22208. PMID 34962526
- [Background] Owolabi MO, Thrift AG, Mahal A, Ishida M, Martins S, Johnson WD, Pandian J, Abd-Allah F, Yaria J, Phan HT, Roth G, Gall SL, Beare R, Phan TG, Mikulik R, Akinyemi RO, Norrving B, Brainin M, Feigin VL; Stroke Experts Collaboration Group. Primary stroke prevention worldwide: translating evidence into action. Lancet Public Health. 2022 Jan;7(1):e74-e85. doi: 10.1016/S2468-2667(21)00230-9. Epub 2021 Oct 29. PMID 34756176